CLINICAL TRIAL: NCT01424891
Title: Effects on NF-κB Activity: High Dose Simvastatin Versus Combination Therapy With Ezetimibe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Gottfried Rudofsky, Principal investigator, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SimEze
Record Dates: First submitted 2011-08-23; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Treatment with placebo over 8 weeks
  Interventions: Drug: Placebo
- Simvastatin 80 mg (Active Comparator): treatment with 80 mg of simvastatin over 8 weeks
  Interventions: Drug: Simvastatin 80 mg
- Sim10/Eze10 (Active Comparator): treatment with 10 mg of simvastatin in combination with 10 mg ezetimibe over 8 weeks
  Interventions: Drug: Sim10/Eze10

INTERVENTIONS:
Drug: Simvastatin 80 mg — treatment with 80 mg of simvastatin over a period of 8 weeks
  Other Names: zocor; simvastatin
  Arms: Simvastatin 80 mg
Drug: Sim10/Eze10 — treatment with combination of simvastatin 10 mg and ezetimibe 10 mg
  Other Names: inegy
  Arms: Sim10/Eze10
Drug: Placebo — treatment with placebo over 8 weeks
  Arms: Placebo

SUMMARY:
Lowering LDL cholesterol by statins has been proven to be associated with reduction of proinflammatory regulators e.g. activation of the transcription factor NF-ĸB. Up to now the effects of newer cholesterol lowering agents such as ezetemibe with respect to their anti-inflammatory potential are less intensively studied. Therefore the investigators analyzed whether equipotent LDL-lowering therapy with simvastatin alone and in combination with ezetimibe have comparable effects on NF-ĸB-activation in peripheral blood mononuclear cells (PBMCs) of patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 80 years old
* type 2 diabetes
* HbA1c value between 6.0 % and 9.0 %
* elevated LDL-c values > 100 mg/dl with no lipid lowering treatment within the last six month

Exclusion Criteria:

* refused informed consent

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-04; Primary Completion 2006-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
NF-kappa B binding activity | up to 5 years
  The binding activity of nuclear transcription factor nuclear factor kappa B (NF-kappa B)will be measured in patients with type 2 diabetes before and after 8 weeks while under study treatment. Analysis will be done with electrophoretic mobility shift assay. Nuclear extract, which is necessary, will be generated from peripheral blood mononuclear cells.

SECONDARY OUTCOMES:
Inflammatory markers | up to 5 years
  Blood levels of high sensitivity CRP and interleukin-6 will be measured before study start and after 8 weeks while under study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Rudofsky, MD, Principal Investigator — University Hospital of Heidelberg
Locations (1):
- University Hospital of Heidelberg, Heidelberg, Germany